CLINICAL TRIAL: NCT04096911
Title: A Single-arm, Single-center, Phase II Clinical Study Evaluating Efficacy of PD-1 Monoclonal Antibody Combined With HPV Vaccine in the Patients With Cervical Cancer（CC）Who Fails in or Can Not Endure the Standard Treatment
Brief Title: Combination of PD-1 Monoclonal Antibody and HPV Vaccine in Patients With Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buhai Wang (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Buhai Wang, doctor, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WBH-7209
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer; Cervical Neoplasms; Cervix Cancer
Keywords: HPV vaccine; PD-1 Monoclonal Antibody; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — sintilimab; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab and HPV Vaccine (Experimental): Sintilimab 200 mg intravenously every 3 weeks ，3 doses of quadrivalent HPV vaccine intramuscularly at day 1,60,180
  Interventions: Drug: Sintilimab; Drug: quadrivalent HPV vaccine

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200 mg intravenously every 3 weeks
  Other Names: IBI308
Drug: quadrivalent HPV vaccine — The first dose of quadrivalent HPV vaccine intramuscularly at the day before the first dose of Sintilimab ，the second and third doses of quadrivalent HPV vaccine intramuscularly at the 60th and 180th days respectively
  Other Names: Gardasil 4

SUMMARY:
The investigators propose to evaluate the efficacy of the combination of Pd-1 Monoclonal Antibody and HPV Vaccine in the patients with cervical cancer who fails in or can not endure the standard treatment

DETAILED DESCRIPTION:
The phase II study is a research which treat cervical carcinoma patients who recurred after at least one prior chemotherapy regimen with Sintilimab and HPV Vaccine. The primary endpoint is objective response rate; secondary endpoints are Progression-Free Survival, Overall Survival and duration of response. Efficacy will be assessed according to RECIST 1.1; progression-free survival is the time from study entry to time of progression or death, whichever occurs first; overall survival is the time from study entry to time of death or the date of last contact,. Furthermore, exploratory studies will be performed on archival tumor material (PD-L1 expression, next-generation sequencing).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have persistent, recurrent or metastatic squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix with documented disease progression (disease not amendable to curative therapy)
2. All patents must have measurable disease as defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam;lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
3. Patients must have at least one "target" lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
4. In the state of HPV infection
5. Appropriate for study entry based on the following diagnostic workup:

   * History/physical examination within 28 days prior to registration
   * Imaging of target lesion(s) within 28 days prior to registration
   * Further protocol-specific assessments:

     * Recovery from adverse effects of recent surgery, radiotherapy or chemotherapy
     * Any other prior therapy directed at the malignant tumor including chemotherapy, biologic/targeted agents and immunologic agents must be discontinued at least three weeks prior to registration Investigation agents must be discontinued for at least 30 days prior to registration
     * Any prior radiation therapy must be completed at least 4 weeks prior to registration
     * At least 4 weeks must have elapsed since any major surgery prior to registration
6. Patients must have had one prior systemic chemotherapeutic regimen for management of persistent, recurrent or metastatic carcinoma of the cervix (e.g.; paclitaxel/cisplatin, paclitaxel/cisplatin/bevacizumab); chemotherapy administered concurrent with primary radiation (e.g.; weekly cisplatin) is not counted as a systemic chemotherapy regimen; adjuvant chemotherapy given following the completion of radiation therapy (or concurrent chemotherapy and radiation therapy) is not counted as a systemic chemotherapy regimen (e.g.; paclitaxel and carboplatin for up to 4 cycles); NOTE: patients who have received more than one prior regimen are NOT eligible
7. Have a performance status of 0 or 1 on the ECOG Performance Scale
8. Absolute neutrophil count (ANC) >= 1,500/ul
9. Platelets >= 100,000/ul
10. Creatinine =< 1.5 x institutional upper limit of normal (ULN) or creatinine clearance (CrCl) >= 40 mL/min using Cockcroft-Gault formula
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN

Exclusion Criteria:

1. Has disease which is amenable to radical treatment with surgery or radiation or a combination of treatments.
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known hypersensitivity to Sintilimab or its formulation
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. History of serotonergic syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 24 months
  complete response plus partial response as determined by RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival | Time from study entry to time of progression or death, whichever occurs first, assessed up to 42 months
  Kaplan-Meier median estimates and curves will be used to describe PFS survival functions
Overall survival | Time from study entry to time of death or the date of last contact, assessed up to 42 months
  Kaplan-Meier median estimates and curves will be used to describe OS survival functions
Duration of Response | Time from the first evaluation of the tumor is CR or PR to the first evaluation is PD or death, assessed up to 42 months
  Kaplan-Meier median estimates and curves will be used to describe DOR survival functions

CONTACTS AND LOCATIONS:
Overall Officials: Buhai Wang, Study Chair — People's hospital of northern jiangsu; Yuechao Wu, Study Director — People's hospital of northern jiangsu
Locations (1):
- People's hospital of northern jiangsu, Yangzhou, Jiangsu, China

REFERENCES:
- [Result] Frenel JS, Le Tourneau C, O'Neil B, Ott PA, Piha-Paul SA, Gomez-Roca C, van Brummelen EMJ, Rugo HS, Thomas S, Saraf S, Rangwala R, Varga A. Safety and Efficacy of Pembrolizumab in Advanced, Programmed Death Ligand 1-Positive Cervical Cancer: Results From the Phase Ib KEYNOTE-028 Trial. J Clin Oncol. 2017 Dec 20;35(36):4035-4041. doi: 10.1200/JCO.2017.74.5471. Epub 2017 Nov 2. PMID 29095678
- [Result] Kranawetter M, Rohrich S, Mullauer L, Obermair H, Reinthaller A, Grimm C, Sturdza A, Kostler WJ, Polterauer S. Activity of Pembrolizumab in Recurrent Cervical Cancer: Case Series and Review of Published Data. Int J Gynecol Cancer. 2018 Jul;28(6):1196-1202. doi: 10.1097/IGC.0000000000001291. PMID 29787422
- [Result] Pembrolizumab OK'd for Cervical Cancer. Cancer Discov. 2018 Aug;8(8):904. doi: 10.1158/2159-8290.CD-NB2018-086. Epub 2018 Jul 2. PMID 29967015
- [Result] Wang Y, Li G. PD-1/PD-L1 blockade in cervical cancer: current studies and perspectives. Front Med. 2019 Aug;13(4):438-450. doi: 10.1007/s11684-018-0674-4. Epub 2019 Mar 2. PMID 30826965
- [Derived] Wang B, Liang Y, Wu Y, Li Q, Zeng Y, Liu L, Cao W, Geng X, Huang Y, Wu Y, Pan J, Zhang X, Gu JJ. Sintilimab plus HPV vaccine for recurrent or metastatic cervical cancer. J Immunother Cancer. 2024 Nov 27;12(11):e009898. doi: 10.1136/jitc-2024-009898. PMID 39608975
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/29095678
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/29787422
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/29967015
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/30826965